CLINICAL TRIAL: NCT05675878
Title: Confirmation of Diet as a Treatment for Gulf War Illness
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: American University (Other)
Collaborators: Boston University (Other); Massachusetts General Hospital (Other); Georgetown University (Other); Nova Southeastern University (Other)
Responsible Party: Principal Investigator, Kathleen Holton, Associate Professor, American University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-46; CDMRP-GW210080 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2022-12-16; First posted 2023-01-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Gulf War Syndrome; Gulf War Illness
Keywords: Gulf War Illness; GWI; Gulf War Syndrome; Diet; Treatment
MeSH Terms: conditions — Persian Gulf Syndrome | interventions — Diet Therapy

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to either immediately start the intervention or to the wait-listed control group. The intervention group will be trained, and then will follow the diet for one month. The waitlisted controls will follow their normal diet for one month, and then will have the opportunity to be trained on the diet and follow the intervention for one month.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary Intervention Group (Experimental): Subjects will undergo a 2-hour in-depth training via Zoom on how to follow the diet and will receive a binder with helpful information. They will be give the weekend to prepare and then will start the diet the following Monday, and will continue following it for 4 weeks before being reassessed in the lab.
  Interventions: Behavioral: Dietary Intervention
- Waitlisted Control Group (No Intervention): The waitlisted control group will follow their usual diet for one month and then will be reassessed (as a comparator group) before being trained on the dietary intervention which they will then follow for the next month.

INTERVENTIONS:
Behavioral: Dietary Intervention — This is a whole food, nutrient-dense diet that aims to remove exposure to specific food additives thought to have negative neurological effects, while also optimizing micronutrient intake.
  Arms: Dietary Intervention Group

SUMMARY:
This clinical trial aims to confirm previous findings from a smaller study which demonstrated significant improvements in all symptoms among veterans with Gulf War Illness after one month on the dietary intervention. The main objectives of this study are: 1) to confirm previous findings of treatment response to the diet in a larger and more diverse group; 2) to examine how changes in the nervous system may be the reason for improvement; and 3) to identify markers which change in the blood after one month on the diet. Participants will have baseline measures collected and then will be randomized into the intervention or wait-listed control group, which they will follow for one month before being reassessed.

DETAILED DESCRIPTION:
The rationale for the proposed research comes from observations from a smaller study which demonstrated profound widespread symptom improvements in veterans with Gulf War Illness (GWI) after one month on the diet. Improvements were noted in every symptom domain and included significant reductions in overall symptom number (with an average of 9 symptoms going away), reduced pain, fatigue, depression, anxiety, and post-traumatic stress disorder (PTSD); and concurrent significant improvements in cognitive function and quality of life. Results also demonstrated that those who improved on the diet had a significant reduction in peripheral inflammation, as compared to those who did not improve on the diet. These benefits have been observed without any negative side effects and the majority of participants continued to follow the diet three months after study completion, suggesting continued improvement and good feasibility. The objectives of this study are: 1) to evaluate whether or not the substantial benefits observed in the recently completed clinical trial hold in a larger group of more diverse veterans with GWI, and 2) to identify blood and/or brain measures which predict improvement on the diet. By recruiting a large group of veterans which are representative of those with GWI, the findings of this research should be applicable to the larger GWI community. The impact of this research could be quite profound, with the diet being a no-risk, low-cost treatment option with no side effects, which allows each individual veteran to take back control of his/her health. There are no direct risks to following the diet since it is a healthy whole-food dietary approach which provides all necessary nutrients. The potential benefits of the diet include improvement in GWI symptoms; improvement in quality of life, potential for improvement in other health markers related to diet (such as obesity, diabetes, cardiovascular disease, high blood pressure) and the possibility of benefit to the larger community. If positive results are confirmed in the proposed study, then the next step would be to teach all Veterans Administration (VA) dietitians how to administer the low glutamate diet so that all veterans have access to it, which should be possible within 1-2 years of the completion of this study.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females of all races and ethnicities who are ≤75 yrs of age
* Served in the 1990-1991 Persian Gulf War
* Fulfill both Center for Disease Control (CDC) and Kansas definitions of Gulf War Illness
* Stable medication regimen for ≥1 month and willing to keep medications and supplements stable throughout study participation

Exclusion Criteria:

* Recent substance use disorder (past year)
* Unwilling to stop using alcohol, tobacco (including vaping) and/or marijuana; or unwilling to change diet
* Diagnosed seizure disorder or severe asthma requiring past hospitalization
* Currently taking medication which affects glutamatergic or GABAergic neurotransmission (but can work with their physician to wean off of these medications prior to participating)

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Total Symptom Score | 1-month
  This measure computes the number of symptoms being experienced in this widespread chronic pain condition, and also computes a score based on severity of each symptom. The raw symptom score ranges from 0-32, and the symptom severity score ranges from 0-96, with higher scores indicative of worse outcomes.
Patient Global Impression of Change Scale (PGIC) | 1-month
  The PGIC is a self-report measure of the amount of change experienced from the treatment using a 7-point scale with the following options: very much worse, much worse, a little worse, no change, a little better, much better, very much better.

SECONDARY OUTCOMES:
McGill Pain Questionnaire | 1-month
  This pain measure inquires about types of pain sensation ranked on a scale of 0 to 3, with a total score from 0-45. Higher scores indicate worse pain.
Chalder Fatigue Score | 1-month
  The Chalder Fatigue Scale measures the extent and severity of fatigue. It is a scale with answers to each question based on both bimodal and likert scores, resulting in a total score of 0-11 and 0-33, with higher scores indicating more fatigue.
Veterans RAND 36 Item Health Survey (VR-36) | 1-month
  This is a 36-item survey used to measure health related quality of life, to estimate disease burden and to evaluate disease-specific impact on general and selected populations. The items on the questionnaire correspond to eight principal health domains including general health perceptions, physical functioning, role limitations due to physical and emotional problems, bodily pain, energy-fatigue, social functioning and mental health. This results in physical and mental health component quality of life scores, each scored from 0-100, with higher scores indicating a better quality of life.
Brief Irritability Questionnaire (BITe) | 1-month
  This short questionnaire assesses anger and irritability with 5 questions ranked on a 6-point scale. Higher scores indicate more irritability.
Center for Epidemiological Studies Depression Scale (CES-D) | 1-month
  This is a 20-item measure that asks individuals to rate how often over the past week they experienced symptoms associated with depression, such as restless sleep, poor appetite, and feeling lonely. Response options range from 0 to 3 for each item (0 = Rarely or None of the Time, 1 = Some or Little of the Time, 2 = Moderately or Much of the time, 3 = Most or Almost All the Time). Scores range from 0 to 60, with high scores indicating greater depressive symptoms.
Generalized Anxiety Disorder Scale (GAD-7) | 1-month
  A brief questionnaire with 7 questions which measure generalized anxiety disorder. The GAD-7 score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of 'not at all', 'several days', 'more than half the days', and 'nearly every day', respectively, and adding together the scores for the seven questions. Total scores range from 0-21, with higher scores indicating more anxiety.
PTSD Checklist for DSM-5 (PCL-5) | 1-month
  The PCL-5 is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. The self-report rating scale is 0-4 for each symptom, reflecting a change from 1-5 in the DSM-IV version. Rating scale descriptors are the same: "Not at all," "A little bit," Moderately," "Quite a bit," and "Extremely." A total symptom severity score (range - 0-80) can be obtained by summing the scores for each of the 20 items, with higher total scores indicating a higher probability of having PTSD.
Cognitive Testing | 1-month
  Cognitive function will be measured using computerized cognitive testing software and one administered exam in-person. An overall score, called a neurocognitive index, is computed as the average of 5 domain scores, with higher scores equating to better cognitive function.
Dolorimetry | 1-month
  Pain threshold will be measured using a dolorimeter, where pressure is applied to 18 points on the body that are typically tender in widespread chronic pain conditions. The participant will report when pain starts and the kilograms of pressure will be recorded. These will be averaged over the 18 sites, with higher scores indicative of having a higher (better) pain threshold.
Biophotonic scanner | 1-month
  A biophotonic scanner will be used to assess long-term carotenoid intake from the diet. This is a painless test where an infared light is shone through the index finger. This results in a numeric score from 0-800, with a higher score indicative of higher dietary carotenoid intake.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen F Holton, PhD, MPH, Principal Investigator — American University
Locations (3):
- United States (3):
  - American University, Washington D.C., District of Columbia
  - Nova Southeastern University, Fort Lauderdale, Florida
  - Boston University, Boston, Massachusetts